CLINICAL TRIAL: NCT02616393
Title: A Phase 2, Multicenter Study of Tesevatinib in Subjects With Non-Small Cell Lung Cancer, EGFR Activating Mutation, Prior Treatment With a Tyrosine Kinase Inhibitor, and Brain Metastases or Leptomeningeal Metastases
Brief Title: Phase 2 Study of Study of Tesevatinib in Subjects With NSCLC and Brain or Leptomeningeal Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD019-206
Record Dates: First submitted 2015-11-20; First posted 2015-11-26 (Estimated); Results first posted 2021-11-23 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Non-Small Cell Lung Cancer; Leptomeningeal Metastases; Brain Metastases
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Meningeal Carcinomatosis; Brain Neoplasms | interventions — XL647

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: Brain Metastases (BM) (Experimental): Tesevatinib 300 mg orally (PO) once daily (QD) administered to subjects with NSCLC who had progressed with brain metastases (BM)
  Interventions: Drug: Tesevatinib
- Cohort B: Leptomeningeal Metastases (LM) (Experimental): Tesevatinib 300 mg PO QD administered to subjects with NSCLC who had progressed with leptomeningeal metastases (LM)
  Interventions: Drug: Tesevatinib
- Cohort C: Brain Metastases at Initial Presentation (BM-IP) (Experimental): Tesevatinib 300 mg PO QD administered NSCLC who presented initially with BM at initial presentation
  Interventions: Drug: Tesevatinib

INTERVENTIONS:
Drug: Tesevatinib
  Other Names: KD019, XL647

SUMMARY:
A study to assess the activity of tesevatinib in subjects with non-small cell lung cancer (NSCLC) and activating epidermal growth factor receptor (EGFR) mutations who have disease progression with Brain Metastases (BM) or Leptomeningeal Metastases (LM) or who have either BM or LM at initial presentation (IP)

DETAILED DESCRIPTION:
This was a multicenter, phase 2, open-label study to assess the activity of tesevatinib, in subjects with non-small cell lung cancer (NSCLC) and activating epidermal growth factor receptor (EGFR) mutations, and brain metastases (BM) or leptomeningeal metastases (LM).

After completion of the screening assessments and confirmation of study eligibility, tesevatinib was orally administered to all subjects at a dose of 300 mg once daily (QD). Tumor response, both in the central nervous system (CNS) and outside the central nervous system (non-CNS), was assessed after the second cycle of treatment and then at the end of every two cycles of treatment thereafter. Subjects were treated with tesevatinib 300 mg QD until disease progression or the subject experienced unacceptable toxicity.

Subjects who discontinued tesevatinib therapy were followed for survival.

Subjects with NSCLC + EGFR mutations were assigned to one of three cohorts:

* Cohort A: Brain Metastases (BM). Subjects had progressed with BM.
* Cohort B: Leptomeningeal Metastases (LM). Subjects had initially presented or progressed with LM.
* Cohort C: Brain Metastases at Initial Presentation (BM-IP). Subjects had no prior systemic therapy.

Each of the three cohorts was to have 20 subjects, for a total of 60 subjects. All three cohorts were enrolled simultaneously.

The primary objectives were to include:

* Clinical activity of tesevatinib of subjects in Cohort A (BM) and Cohort C (BM-IP) as measured by Response Criteria in Solid Tumors (RECIST) version 1.1 which evaluated changes in BM size.
* Clinical activity of tesevatinib of subjects in Cohort B (LM) as measured by improvement in Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 symptoms and signs.

Efficacy assessments included response to treatment using RECIST criteria, progression-free survival (PFS), time to progression (TTP), overall survival (OS), and Quality of Life (QOL) questionnaires. Safety assessments included adverse event (AE) monitoring, electrocardiogram (ECG), Eastern Cooperative Oncology Group (ECOG) Performance Status, laboratory testing, physical examination, vital signs, and pregnancy testing. In addition, pharmacokinetic (PK) and pharmacodynamic (PD) assessments were performed.

An End of Treatment Visit occurred within 3 days after the subject's last dose of study drug. This could have occurred at the visit when disease progression was diagnosed. Subjects were continued to be followed for disease progression and survival.

A follow-up visit occurred 30 days (± 5 days) after the last dose of study drug. This visit may have occurred prior to 30 days if a new therapy was started within 30 days of last dose of study drug.

For long-term follow-up, after subjects withdrew from the active treatment portion of the study, they were contacted by telephone every 8 weeks to assess survival status and any subsequent anti-cancer treatment.

ELIGIBILITY:
Cohort A

Inclusion Criteria:

* History of non-small cell lung cancer (NSCLC) with epidermal growth factor receptor (EGFR) mutation or an EGFR activating mutation that has had a clinical response to erlotinib, afatinib, or gefitinib in the patient being enrolled
* Occurrence or progression of BM while receiving first-line therapy (either erlotinib, afatinib, or gefitinib) for at least 14 days. Patients may have received osimertinib (or other agents inhibiting the T790M EGFR mutation) as second line therapy. If BM progression occurs after osimertinib, patient will be eligible.
* At least one measurable BM by RECIST 1.1 criteria (≥ 10 mm in longest diameter). Target lesions must not have received stereotactic radiotherapy (SRS). If a subject had prior whole brain radiotherapy (WBRT), progression in any measurable BM lesion must have occurred at least 3 months after the end of WBRT. Subjects with asymptomatic brain metastases may have been enrolled without prior radiation therapy to the brain. Subjects with minimally symptomatic brain metastases may have been enrolled without prior radiation therapy to the brain if they do not require immediate surgical or radiation therapy in the opinion of the treating investigator and in the opinion of a radiation therapy or neurosurgical consultant
* Subjects in Cohort A may have had asymptomatic LM detected by MRI. (Subjects with symptoms or signs attributed to LM were enrolled in Cohort B whether or not they have brain metastases)
* No clinically significant progression outside of the CNS on most recent EGFR inhibitor therapy
* ECOG Score ≤ 2
* No history of another malignancy in the 5 years prior to study entry, except treated non-melanoma skin cancer or superficial bladder cancer or carcinoma in situ of the cervix or Stage 1 or 2 cancers of other sites that have been treated surgically and have not recurred
* Adequate organ and bone marrow functions
* Serum potassium and magnesium levels above the lower limit of normal
* No coexisting medical problems of sufficient severity to limit compliance with the study
* Willing and able to sign written informed consent and able to comply with the study protocol for the duration of the study
* Women of childbearing potential (i.e., menstruating women) must have had a negative urine pregnancy test (positive urine tests confirmed by serum test)

Exclusion Criteria:

* First day of dosing with tesevatinib less than 2 weeks from the last treatment of cytotoxic chemotherapy, biological therapy, or immunotherapy, and less than 6 weeks for nitrosoureas and mitomycin C. Surgical procedures must have been performed at least 2 weeks prior to the start of study treatment. Subjects must have recovered from the reversible effects of prior lung cancer treatments, including surgery and radiation therapy (excluding alopecia).
* First day of dosing with tesevatinib less than 4 weeks from the last radiotherapy of the brain or spinal cord/cauda equina
* First day of dosing with tesevatinib less than 2 weeks from treatment with another investigational agent
* Treatment with erlotinib must have been discontinued at least 3 days prior to first dose of tesevatinib and treatment with afatinib or other tyrosine kinase inhibitor must have been discontinued at least 3 days prior to first dose of tesevatinib
* Any concurrent therapy for BM other than the specified treatment in this study
* Taking any medication known to moderately or severely inhibit the CYP3A4 isozyme or any drugs that are CYP3A4 inducers (including anti-epileptic agents such as phenytoin). A stable regimen (≥ 4 weeks) of antidepressants of the selective serotonin uptake inhibitor (SSRI) class was allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline, and fluoxetine)
* Taking any drugs associated with torsades de pointes or known to moderately or severely prolong the QTc(F) interval
* Evidence of active heart disease such as myocardial infarction within the 3 months prior to study entry; symptomatic coronary insufficiency congestive heart failure; moderate or severe pulmonary dysfunction
* History of torsades de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first degree block, being PR interval only), or congenital long QT syndrome. Subjects with a history of atrial arrhythmias were discussed with the medical monitor
* Had an active infectious process
* Female subject pregnant or lactating
* Known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Marked prolongation of QTc(F) interval at screening or baseline (QTc[F] interval > 470 msec) using the Fridericia method of correction for heart rate
* Gastrointestinal (GI) condition interfering with drug absorption
* Non-malignant neurological disease that would interfere with evaluation of symptoms or signs of brain metastases

Cohort B

Inclusion Criteria:

* History of NSCLC with EGFR mutation (either exon 19 deletion or L858R mutation) or, if previously treated, history of an activating EGFR mutation that had a clinical response to erlotinib, afatinib, or gefitinib in the subject being enrolled).
* Presentation with LM at initial presentation with no prior systemic treatment, or occurrence or progression of LM while receiving first-line therapy (either erlotinib, afatinib, or gefitinib) for at least 14 days. Patients may have received osimertinib (or other agents inhibiting the T790M EGFR mutation) as second line therapy. If LM progression occurred after osimertinib, subjects were eligible.
* Presence of at least one CTCAE 4.03 symptom/sign of at least Grade 1 attributed by the investigator to LM
* Diagnosis of LM by:

  1. Cytological evidence in cerebrospinal fluid (CSF) sample of LM due to NSCLC, and/or
  2. Findings on gadolinium-enhanced MRI
* No clinically significant progression outside of the CNS on most recent EGFR inhibitor therapy
* Concomitant brain metastases and brain metastases previously treated with radiation therapy were allowed. (Subjects with symptoms or signs attributed to LM will be enrolled in Cohort B whether or not they have brain metastases)
* ECOG Score ≤ 2
* No history of another malignancy in the 5 years prior to study entry, except treated non-melanoma skin cancer or superficial bladder cancer or carcinoma in situ of the cervix or Stage 1 or 2 cancers of other sites that have been treated surgically and had not recurred
* Adequate organ and bone marrow functions
* Serum potassium and magnesium levels above the lower limit of normal (LLN)
* No coexisting medical problems of sufficient severity to limit compliance with the study
* Willing and able to sign written informed consent and able to comply with the study protocol for the duration of the study
* Women of childbearing potential (i.e., menstruating women) must have had a negative urine pregnancy test (positive urine tests confirmed by serum test)

Exclusion Criteria:

* First day of dosing with tesevatinib less than 2 weeks from the last treatment of cytotoxic chemotherapy, biological therapy, or immunotherapy, and less than 6 weeks for nitrosoureas and mitomycin C. Surgical procedures must have been performed at least 2 weeks prior to the start of study treatment. Subjects must have recovered from the reversible effects of prior lung cancer treatments, including surgery and radiation therapy (excluding alopecia).
* First day of dosing with tesevatinib less than 4 weeks from the last radiotherapy of the brain or spinal cord/cauda equina
* First day of dosing with tesevatinib less than 2 weeks from treatment with another investigational agent
* Treatment with erlotinib must have been discontinued at least 3 days prior to first dose of tesevatinib and treatment with afatinib or other tyrosine kinase inhibitor must have been discontinued at least 3 days prior to first dose of tesevatinib
* Any concurrent therapy for LM other than the specified treatment in this study
* Taking any medication known to moderately or severely inhibit the CYP3A4 isozyme or any drugs that are CYP3A4 inducers (including anti-epileptic agents such as phenytoin). A stable regimen (≥ 4 weeks) of antidepressants of the SSRI class was allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline, and fluoxetine)
* Taking any drugs associated with torsades de pointes or known to moderately or severely prolong the QTc(F) interval
* Evidence of active heart disease such as myocardial infarction within the 3 months prior to study entry; symptomatic coronary insufficiency congestive heart failure; moderate or severe pulmonary dysfunction
* History of torsades de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first degree block, being PR interval only), or congenital long QT syndrome. Subjects with a history of atrial arrhythmias were discussed with the medical monitor.
* Has an active infectious process
* Female subject pregnant or lactating
* Known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Marked prolongation of QTc(F) interval at screening or baseline (QTc[F] interval > 470 msec) using the Fridericia method of correction for heart rate
* GI condition that would interfere with drug absorption
* Non-malignant neurological disease that would interfere with evaluation of symptoms or signs of leptomeningeal metastases
* Contraindications to lumbar puncture:

  1. International Normalized Ratio (INR) > 1.5
  2. Platelets < 50 × 10^9/L (Note that platelets are required to be ≥100× 10^9/L at screening)
  3. Therapeutic anticoagulant treatment that can't be held for 24 hours. Low dose low molecular weight heparin given for deep vein thrombosis (DVT) prophylaxis was allowed.
  4. CNS lesions considered to be at risk for cerebral herniation, myelocompression, or conus/cauda compression

Cohort C

Inclusion Criteria:

* NSCLC with EGFR activating mutation
* No prior systemic treatment for NSCLC. Treatment with systemic steroids was not considered systemic treatment for NSCLC
* No prior radiation therapy to the CNS (brain or spinal cord)
* At least one measurable BM by RECIST 1.1 criteria (≥ 10 mm in longest diameter) in a subject with asymptomatic or minimally symptomatic brain metastases who did not require immediate surgical or radiation therapy in the opinion of the treating investigator and in the opinion of a radiation therapy or neurosurgical consultant.
* Subjects in Cohort C may have had asymptomatic LM detected by MRI
* ECOG Score ≤ 2
* No history of another malignancy in the 5 years prior to study entry, except treated non-melanoma skin cancer or superficial bladder cancer or carcinoma in situ of the cervix or Stage 1 or 2 cancers of other sites that have been treated surgically and have not recurred
* Adequate organ and bone marrow functions
* Serum potassium and magnesium levels above the LLN
* No coexisting medical problems of sufficient severity to limit compliance with the study.
* Willing and able to sign written informed consent and able to comply with the study protocol for the duration of the study
* Women of childbearing potential (i.e., menstruating women) must have had a negative urine pregnancy test (positive urine tests are to be confirmed by serum test)

Exclusion Criteria:

* Surgical procedures performed less than 2 weeks prior to the start of study treatment
* Any concurrent therapy for BM other than the specified treatment in this study
* Taking any medication known to moderately or severely inhibit the CYP3A4 isozyme or any drugs that are CYP3A4 inducers (including anti-epileptic agents such as phenytoin). A stable regimen (≥ 4 weeks) of antidepressants of the SSRI class was allowed (common SSRIs include escitalopram oxalate, citalopram, fluvoxamine, paroxetine, sertraline, and fluoxetine)
* Taking any drugs associated with torsades de pointes or known to moderately or severely prolong the QTc(F) interval
* Evidence of active heart disease such as myocardial infarction within the 3 months prior to study entry; symptomatic coronary insufficiency congestive heart failure; moderate or severe pulmonary dysfunction
* History of torsades de pointes, ventricular tachycardia or fibrillation, pathologic sinus bradycardia (< 50 bpm), heart block (excluding first-degree block, being PR interval only), or congenital long QT syndrome. Subjects with a history of atrial arrhythmias were discussed with the medical monitor
* An active infectious process
* Female subject pregnant or lactating
* Known contraindication to MRI, such as cardiac pacemaker, shrapnel, or ocular foreign body
* Marked prolongation of QTc(F) interval at screening or Cycle 1 Day 1 (QTc[F] interval > 470 msec) using the Fridericia method of correction for heart rate
* GI condition interfering with drug absorption
* Non-malignant neurological disease that would interfere with evaluation of symptoms or signs of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-11; Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - USC Norris Oncology/Hematology Newport Beach, Newport Beach, California
  - John Wayne Cancer Institute, Santa Monica, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UT M.D. Anderson Cancer Center, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A (BM): Subjects with brain metastases (BM) who received tesevatinib 300 mg orally (PO) once daily (QD)
- Cohort B (LM): Subjects with leptomeningeal metastases (LM) who received tesevatinib 300 mg PO QD
- Cohort C (BM-IP): Subjects with brain metastases at initial presentation (BM-IP) who received tesevatinib 300 mg PO QD
Period: Overall Study
Arm/Group | Cohort A (BM) | Cohort B (LM) | Cohort C (BM-IP)
Started | 13 | 20 | 3
Completed | 0 | 0 | 0
Not Completed | 13 | 20 | 3
Not completed — Death | 5 | 12 | 1
Not completed — Termination by Sponsor | 4 | 5 | 2
Not completed — Other | 3 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Lost to Follow-up | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort A - Brain Metastases: Tesevatinib will be orally administered with a dose of 300 mg once daily to subjects with NSCLC who have progressed with BM
  Tesevatinib
- Cohort B - Leptomeningeal Metastases: Tesevatinib will be orally administered with a dose of 300 mg once daily to subjects with NSCLC who have progressed with LM
  Tesevatinib
- Cohort C - Brain Metastases at Initial Presentation: Tesevatinib will be orally administered with a dose of 300 mg once daily to subjects with NSCLC with BM at initial presentation
  Tesevatinib
- Total: Total of all reporting groups
Arm/Group | Cohort A - Brain Metastases | Cohort B - Leptomeningeal Metastases | Cohort C - Brain Metastases at Initial Presentation | Total
Number analyzed (Participants) | 13 | 20 | 3 | 36
Age, Continuous [Mean (Full Range); unit: years] | 60.7 [50.0 to 77.0] | 56.3 [36.0 to 82.0] | 64.7 [57.0 to 82.0] | 58.6 [36.0 to 82.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 15 | 2 | 23
  Male | 7 | 5 | 1 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 10 | 19 | 3 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 3 | 10 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 2 | 6
  White | 4 | 8 | 1 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 4 | 0 | 0 | 4
EORTC-QLQ-C30 Questionnaire [Mean (Standard Deviation); unit: Units (score) on a scale] — The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer 30 (C30) is 30-question assessment scales: 5 functional; 3 symptom; 1 global QoL scale and, 6 single items; rated on 4-point scale (not at all, a little, quite a bit, very much) scored 0 to 100. High score for functional scale = high/healthy functioning; high score for global health = high QoL; but high score for symptom scale = high level of symptomatology/problems.
  Units (score) on a scale | 59.2 (20.48) | 66.5 (12.84) | 51.7 (5.51) | 62.7 (60.6)
EORTC-QLQ-BN20 Questionnaire [Mean (Standard Deviation); unit: Units (score) on a scale] — The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer BN20 Questionnaire is a 20-question assessment of symptomatology based on a categorical scale (Not at all = 1; A little = 2; Quite a bit = 3; and Very much = 4). For 20 questions: minimum score = 20 and maximum score = 80. Higher scores indicate greater level of symptomatology/problems.
  Units (score) on a scale | 34.0 (15.71) | 37.7 (8.64) | 22.0 (2.00) | 35.1 (11.89)

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR) of Subjects With BM
Description: The best overall response rates (ORRs) of subjects who had brain tumors and exhibited either a complete response (CR) or a partial responder (PR) to therapy divided by the total number of subjects treated with tesevatinib 300 mg PO QD. Response rates are in accordance with RECIST Version 1.1 criteria. Since such brain metastases (BM) tumors can either affect the central nervous system (CNS) or not affect the CNS (non-CNS), they were categorized into CNS and non-CNS subsets. Because leptomeningeal metastases (LM) only are considered cancer cell migration from the breast, lung, or some other part of the body to the cerebrospinal fluid (CSF), analysis of CNS are not appropriate, so Cohort B is excluded.
Time Frame: Until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first
Population: Subjects with BM only (Cohorts A and C). Subjects with LM (Cohort B) were excluded.
Measure: Number (95% Confidence Interval); unit: Percentage of participants (%)
Groups:
- Overall BM: All subjects with brain metastases who received tesevatinib 300 mg PO QD
Arm/Group | Cohort A (BM) | Cohort C (BM-IP) | Overall BM
Number analyzed (Participants) | 13 | 3 | 16
Percentage of participants (%)
  CNS | 15.4 [2 to 45] | 100 [29 to 100] | 31.3 [11 to 59]
  non-CNS | 0 [0 to 25] | 100 [29 to 100] | 18.8 [4 to 46]
  CNS + non-CNS | 15.4 [2 to 45] | 100 [29 to 100] | 31.3 [11 to 59]

2. Primary Outcome: Best ORR of Subjects With LM
Description: The best overall response rates (ORRs) of subjects who had leptomeningeal tumors and exhibited either a complete response (CR) or a partial responder (PR) to therapy divided by the total number of subjects treated with tesevatinib 300 mg PO QD. Response rates are in accordance with RECIST Version 1.1 criteria. Since leptomeningeal metastases (LM) are only considered cancer cell migration from the breast, lung, or some other part of the body to the cerebrospinal fluid (CSF), analysis of CNS are not appropriate, so Cohorts A and C are excluded.
Time Frame: Until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first
Measure: Number; unit: Percentage of participants (%)
Groups:
- Cohort B (LM): Subjects with leptomeningeal metastases (LM) who received 300 mg PO QD
Arm/Group | Cohort B (LM)
Number analyzed (Participants) | 20
Percentage of participants (%) | 0

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Median duration of survival without progression of subjects treated with tesevatinib 300 mg PO QD.
Time Frame: Until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Cohort A (BM): Subjects with brain metastases (BM) administered tesevatinib 300 mg orally (PO) once daily (QD)
- Cohort B (LM): Subjects with leptomeningeal metastases (LM) administered tesevatinib 300 mg orally (PO) once daily (QD)
- Cohort C (BM-IP): Subjects with brain metastases at initial presentation (BM-IP) administered tesevatinib 300 mg orally (PO) once daily (QD)
Arm/Group | Cohort A (BM) | Cohort B (LM) | Cohort C (BM-IP)
Number analyzed (Participants) | 13 | 20 | 3
Weeks | 9.29 [4.14 to 27.43] | 10.86 [6.86 to 17.14] | 37.71 [20.14 to 62.14]

4. Secondary Outcome: Probability of PFS at 12 Weeks and 24 Weeks--Cohort A (BM Only) and Cohort B (LM Only)
Description: Probability that subjects with brain metastases (BM) or leptomeningeal metastases (LM) would not progress, i.e., progression-free survival (PFS) after 12 weeks (3 months) and after 24 weeks (6 months) of treatment with tesevatinib 300 mg PO QD
Time Frame: 24 weeks (6 months)
Population: Note: Cohort C (BM-IP) did not have a sufficient number of subjects with events to determine the PFS at 12 or 24 weeks.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Cohort A (BM) | Cohort B (LM)
Number analyzed (Participants) | 13 | 20
Probability
  12 weeks (3 months) | 0.4762 [0.1823 to 0.7237] | 0.4737 [0.2444 to 0.6728]
  24 weeks (6 months) | 0.2857 [0.0698 to 0.5546] | 0.2632 [0.0958 to 0.4677]

5. Secondary Outcome: Probability of PFS at 24 Weeks--Cohort C (BM-IP Only)
Description: Probability that subjects with brain metastases at initial presentation (BM-IP) would not progress, i.e., progression-free survival (PFS) after 24 weeks (6 months) of treatment with tesevatinib 300 mg PO QD
Time Frame: 24 weeks (6 months)
Population: Note: Insufficient data for PFS probability at 12 weeks
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Cohort C (BM-IP)
Number analyzed (Participants) | 3
Probability | 0.6667 [0.0541 to 0.9452]

6. Secondary Outcome: Probability of OS at 12 Weeks and at 24 Weeks--Cohort A (BM Only) and Cohort B (LM Only)
Description: Probability that subjects with brain metastases (BM) or leptomeningeal metastases (LM) survived (overall survival [OS]) after 12 weeks (3 months) and after 24 weeks (6 months) of treatment with tesevatinib 300 mg PO QD
Time Frame: 24 weeks (6 months)
Population: Note: Cohort C did not have a sufficient number of subjects with events to determine the probability of survival at 12 or 24 weeks.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Cohort A (BM) | Cohort B (LM)
Number analyzed (Participants) | 13 | 20
Probability
  12 weeks (3 months) | 0.8462 [0.5122 to 0.9591] | 0.8471 [0.5968 to 0.9480]
  24 weeks (6 months) | 0.7692 [0.4421 to 0.9191] | 0.6353 [0.3831 to 0.8070]

7. Secondary Outcome: Median Time to Progression (TTP)--Cohort A (BM), Cohort B (LM), Cohort C (BM-IP)
Description: Median time to the development of disease progression (TTP) for subjects in Cohort A, Cohort B and Cohort C who were treated with tesevatinib 300 mg PO QD
Time Frame: Until disease progression, death, unacceptable toxicity, or up to 2 years, whichever occurred first
Measure: Median (95% Confidence Interval); unit: Weeks
Groups:
- Cohort B (LM): Subjects with leptomeningeal metastases (LM) who were administered tesevatinib 300 mg orally (PO) once daily (QD)
- Cohort C (BM-IP): Subjects with brain metastases at initial presentation who were administered 300 mg PO QD
Arm/Group | Cohort A (BM) | Cohort B (LM) | Cohort C (BM-IP)
Number analyzed (Participants) | 13 | 20 | 3
Weeks | 21.43 [4.14 to 27.43] | 8.14 [6.00 to 35.86] | 34.93 [32.14 to 37.71]

8. Secondary Outcome: Probability of TTP at 12 Weeks and 24 Weeks--Non-CNS Cohort A (BM Only) and Cohort B (LM Only)
Description: Probability that the time to progression (TTP) for subjects with no metastases to the central nervous system (non-CNS) in Cohort A (brain metastases only) or Cohort B (leptomeningeal metastases only) would be at 12 weeks (3 months) and at 24 weeks (6 months) of therapy with tesevatinib 300 mg PO QD. There were an insufficient number of subjects in Cohort C (brain metastases at initial presentation) who had events.
Time Frame: 24 weeks (6 months)
Population: Note: Cohort C (BM-IP) did not have a sufficient number of subjects with events to determine the probability of TTP at 12 weeks or 24 weeks.
Measure: Number (95% Confidence Interval); unit: Probability
Arm/Group | Cohort A (BM) | Cohort B (LM)
Number analyzed (Participants) | 13 | 20
Probability
  Non-CNS at 12 weeks | 0.5625 [0.1468 to 0.8415] | 0.4396 [0.1684 to 0.6844]
  Non-CNS at 24 weeks | 0.2813 [0.0135 to 0.6880] | 0.2637 [0.0650 to 0.5521]

9. Secondary Outcome: Probability of TTP at 24 Weeks--CNS
Description: Probability that the time to progression (TTP) for subjects with metastases to the central nervous system (CNS) would be at 24 weeks (6 months) of therapy with tesevatinib 300 mg PO QD.
Time Frame: 24 weeks (6 months)
Measure: Number (95% Confidence Interval); unit: Probability
Groups:
- Cohort A - Brain Metastases: Tesevatinib administered at a dose of 300 mg PO QD to subjects with NSCLC who progressed with BM
- Cohort B - Leptomeningeal Metastases: Tesevatinib administered at a dose of 300 mg PO QD to subjects with NSCLC who progressed with LM
- Cohort C - Brain Metastases at Initial Presentation: Tesevatinib administered at a dose of 300 mg PO QD to subjects with NSCLC with BM at initial presentation
Arm/Group | Cohort A - Brain Metastases | Cohort B - Leptomeningeal Metastases | Cohort C - Brain Metastases at Initial Presentation
Number analyzed (Participants) | 13 | 20 | 3
Probability | 0.3636 [0.0584 to 0.6976] | 0.4795 [0.1541 to 0.7491] | 0.5000 [0.0060 to 0.9104]

10. Secondary Outcome: Quality of Life (QoL): Mean Change From Baseline in EORTC-QLQ-C30 Questionnaire Scores
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer 30 (C30) is a 30-question assessment composed of both multi-item scales and single-item measures: 5 functional scales, 3 symptom scales, 1 global QoL scale, and 6 single items. Ratings are on a 4-point scale (not at all, a little quite a bit, very much), with scoring from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning, a high score for the global health status/QoL represents a high QoL, but a high score for a symptom scale/item represents a high level of symptomatology/problems. The outcome measure is the mean change in the EORTC-QLQ-C30 from baseline to a visit.
Time Frame: Until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first
Population: Note: Not all subjects were available for analysis at all visits.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Cohort A (BM): Subjects with brain metastases (BM) who were administered tesevatinib 300 mg orally (PO) once daily (QD)
- Cohort B (LM): Subjects with leptomeningeal metastases (LM) who were administered tesevatinib 300 mg PO QD
- Cohort C (BM-IP): Subjects with brain metastases at initial presentation (BM-IP) who were administered tesevatinib 300 mg PO QD
- All Subjects (Cohorts A+B+C): All subjects with BM, LM or BM-IP who were administered tesevatinib 300 mg PO QD
Arm/Group | Cohort A (BM) | Cohort B (LM) | Cohort C (BM-IP) | All Subjects (Cohorts A+B+C)
Number analyzed (Participants) | 13 | 20 | 3 | 36
Score on a scale
  Baseline Score (35 subjects): number analyzed (Participants) | 12 | 20 | 3 | 35
  Baseline Score (35 subjects) | 59.2 (20.48) | 66.5 (12.84) | 51.7 (5.51) | 62.7 (15.91)
  Mean Change--Cycle 3 Day 1 Change From Baseline: number analyzed (Participants) | 7 | 9 | 3 | 19
  Mean Change--Cycle 3 Day 1 Change From Baseline | 3.6 (5.22) | 2.1 (12.09) | 3.3 (0.58) | 2.8 (8.64)
  Mean Change from Baseline--Cycle 5 Day 1: number analyzed (Participants) | 5 | 2 | 3 | 10
  Mean Change from Baseline--Cycle 5 Day 1 | 2.8 (4.21) | 5.5 (10.61) | 1.0 (5.00) | 2.8 (5.35)
  Mean Change from Baseline to End-of-Study: number analyzed (Participants) | 8 | 9 | 3 | 20
  Mean Change from Baseline to End-of-Study | 2.9 (5.17) | 7.2 (14.34) | 15.0 (4.00) | 6.7 (10.74)

11. Secondary Outcome: Quality of Life (QoL): Mean Change From Baseline in EORTC-QLQ-BN20 Questionnaire Scores
Description: The European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) Cancer BN20 Questionnaire is a 20-question assessment of symptomatology based on a categorical scale (Not at all = 1; A little = 2; Quite a bit = 3; and Very much = 4). For 20 questions: minimum score = 20 and maximum score = 80. Higher scores indicate greater level of symptomatology/problems. The outcome measure is the mean change in the EORTC-QLQ-BN20 from baseline to a visit.
Time Frame: Until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first
Population: Not all subjects were available for all analyses.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Cohort A (BM) | Cohort B (LM) | Cohort C (BM-IP) | All Subjects (Cohorts A+B+C)
Number analyzed (Participants) | 13 | 20 | 3 | 36
Score on a scale
  Baseline Score (35 subjects): number analyzed (Participants) | 12 | 20 | 3 | 35
  Baseline Score (35 subjects) | 34.0 (15.71) | 37.7 (8.64) | 22.0 (2.00) | 35.1 (11.89)
  Mean Change from Baseline--Cycle 3 Day 1 Change From Baseline: number analyzed (Participants) | 7 | 9 | 3 | 19
  Mean Change from Baseline--Cycle 3 Day 1 Change From Baseline | 0.3 (4.89) | 1.9 (6.66) | 3.7 (2.08) | 1.6 (5.44)
  Mean Change from Baseline--Cycle 5 Day 1 Change From Baseline: number analyzed (Participants) | 5 | 2 | 3 | 10
  Mean Change from Baseline--Cycle 5 Day 1 Change From Baseline | -4.0 (5.34) | 2.5 (12.02) | 8.7 (8.96) | 1.1 (8.97)
  Mean Change from Baseline to End-of-Study: number analyzed (Participants) | 7 | 9 | 3 | 19
  Mean Change from Baseline to End-of-Study | 2.6 (3.05) | 7.3 (12.35) | 12.3 (10.26) | 6.4 (9.73)

ADVERSE EVENTS:
Time Frame: Subjects were treated with tesevatinib 300 mg QD until disease progression, unacceptable toxicity, or up to 2 years, whichever occurred first.
Groups:
- Cohort A - Brain Metastases: Tesevatinib 300 mg administered orally (PO) once daily (QD) to subjects with NSCLC who have progressed with BM
- Cohort B - Leptomeningeal Metastases: Tesevatinib 300 mg administered PO to subjects with NSCLC who have progressed with LM
- Cohort C - Brain Metastases at Initial Presentation: Tesevatinib 300 mg administered PO to subjects with NSCLC who presented initially with brain metastases
- All Subjects (Cohorts A+B+C): Tesevatinib 300 mg administered PO to all subjects with NSCLC who had brain metastases and who had leptomeningeal metastases
Arm/Group | Cohort A - Brain Metastases | Cohort B - Leptomeningeal Metastases | Cohort C - Brain Metastases at Initial Presentation | All Subjects (Cohorts A+B+C)
All-Cause Mortality (participants affected / at risk) | 5/13 | 12/20 | 1/3 | 18/36
Serious Adverse Events (participants affected / at risk) | 6/13 | 13/20 | 2/3 | 21/36
Other Adverse Events (participants affected / at risk) | 13/13 | 20/20 | 3/3 | 36/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Brain Metastases (N=13) | Cohort B - Leptomeningeal Metastases (N=20) | Cohort C - Brain Metastases at Initial Presentation (N=3) | All Subjects (Cohorts A+B+C) (N=36)
Urinary tract infection (Infections and infestations) | 1 | 2 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
Disease progression (General disorders) | 0 | 1 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 1
Gait disturbance (General disorders) | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 0 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pneumonthorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 1 | 0 | 1
Subdural hematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - Brain Metastases (N=13) | Cohort B - Leptomeningeal Metastases (N=20) | Cohort C - Brain Metastases at Initial Presentation (N=3) | All Subjects (Cohorts A+B+C) (N=36)
Diarrhea (Gastrointestinal disorders) | 10 | 14 | 0 | 24
Fatigue (General disorders) | 5 | 8 | 3 | 16
QT Prolongation (Investigations) | 5 | 9 | 1 | 15
Nausea (General disorders) | 7 | 5 | 1 | 36
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 3 | 11
Urinary tract infection (Infections and infestations) | 4 | 5 | 1 | 10
Vomiting (Gastrointestinal disorders) | 3 | 5 | 1 | 9
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 3 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1 | 7
Headache (Nervous system disorders) | 2 | 5 | 0 | 7
Hypokalemia (Metabolism and nutrition disorders) | 1 | 4 | 1 | 6
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2 | 5
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0 | 5
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 4 | 0 | 5
Dizziness (Nervous system disorders) | 1 | 2 | 2 | 5
Dysarthria (Nervous system disorders) | 0 | 5 | 0 | 5
Fall (Injury, poisoning and procedural complications) | 2 | 3 | 0 | 5
Gait disturbance (General disorders) | 2 | 3 | 0 | 5
Hypertension (Vascular disorders) | 3 | 2 | 0 | 5
Paresthesia (Nervous system disorders) | 3 | 2 | 0 | 5
Alanine aminotransaminase (ALT) increased (Investigations) | 1 | 3 | 0 | 4
Anal incontinence (Gastrointestinal disorders) | 1 | 3 | 0 | 4
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 4
Dysphagia (Gastrointestinal disorders) | 0 | 4 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 3
Aspartate aminotransferase (AST) increased (Investigations) | 2 | 1 | 0 | 3
Bradycardia (Cardiac disorders) | 2 | 0 | 1 | 3
Confusional state (Psychiatric disorders) | 1 | 2 | 0 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 3
Dysgeusia (Nervous system disorders) | 0 | 1 | 2 | 3
Neuropathy peripheral (Nervous system disorders) | 0 | 2 | 1 | 3
Upper respiratory infection (Infections and infestations) | 1 | 2 | 0 | 3
Urinary retention (Renal and urinary disorders) | 1 | 2 | 0 | 3
Weight decreased (Investigations) | 2 | 1 | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 2 | 2
Asthenia (General disorders) | 1 | 1 | 0 | 2
Balance disorder (Nervous system disorders) | 0 | 2 | 0 | 2
Blood creatinine increased (Investigations) | 1 | 1 | 0 | 2
Chest discomfort (General disorders) | 1 | 1 | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Diplopia (Eye disorders) | 0 | 2 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 2
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Encephalopathy (Nervous system disorders) | 0 | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2
Facial paresis (Nervous system disorders) | 0 | 2 | 0 | 2
Failure to thrive (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hypoesthesia (Nervous system disorders) | 0 | 1 | 1 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hypotension (Vascular disorders) | 1 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 2
Lipase increased (Investigations) | 1 | 1 | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Edema peripheral (General disorders) | 2 | 0 | 0 | 2
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 2
Peripheral swelling (General disorders) | 1 | 1 | 0 | 2
Proteinuria (Renal and urinary disorders) | 2 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 2
Seizure (Nervous system disorders) | 1 | 1 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0 | 2
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0 | 2
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Vision blurred (Eye disorders) | 0 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/93/NCT02616393/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02616393/SAP_001.pdf